CLINICAL TRIAL: NCT05759325
Title: Application of ctDNA-MRD in the Prediction of Curative Effect, Recurrence Monitoring and Prognosis Evaluation of Esophageal Squamous Cell Carcinoma (ESCC) During Perioperative Treatment
Brief Title: An Exploratory Study of ctDNA-MRD in Predicting the Efficacy of Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Jun Liu, GuangzhouIRD, Guangzhou Institute of Respiratory Disease
Other Study IDs: ESCC ctDNA-MRD
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Squamous Cell Carcinoma of Esophagus
Keywords: ESCC; ctDNA
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood before and after surgery, 2 weeks after the end of adjuvant treatment, follow-up period (every 3 months if there is no postoperative treatment), the progress of the disease, as well as the pathological tissues of the initial diagnosis puncture or surgical resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to observe and evaluate the correlation between ctDNA-MRD and the therapeutic effect and prognosis of stage II-IVA operable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
ESCC patients with II-IVA resection will undergo MRD examination at the following time: the first examination is before the operation, the second examination is 7-10 days after the operation, and then 1 month after the operation, 2 weeks after the end of adjuvant treatment (if available), the follow-up period (every 3 months if there is no postoperative treatment) and the progress (the progress of the disease confirmed by the researcher), the patients will receive close MRD monitoring to evaluate the correlation between ctDNA-MRD and therapeutic efficacy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage II-IVA Esophageal squamous cell carcinoma confirmed by clinical pathological staging;
2. ≥18 years;
3. Eastern Cooperative Oncology Group performance status score (ECOG PS) is 0 ~ 1 points;
4. Expected survival time ≥ 6 months;
5. Patients agree and have the ability to follow the planned study visits, laboratory tests and other research steps.

Exclusion Criteria:

1. Patients with other malignant tumors;
2. Patient had undergone surgery before admission;
3. Pregnant or lactating women;
4. Patients with other serious diseases;
5. Patients who could not understand the experiment content and could not cooperate with them and refused to sign the informed consent form;
6. Patients with contraindications to radiotherapy and chemotherapy;
7. Other researchers think it is not suitable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal squamous cell carcinoma patients who were initially diagnosed as stage II-IVA (TNM V8) and planned to undergo radical surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 2 year
  Evaluation of progression-free survival rate of esophageal squamous cell carcinoma patients with different MRD status during perioperative period